CLINICAL TRIAL: NCT03596723
Title: Safety and Efficacy of KPI-121 1% Ophthalmic Suspension Versus Prednisolone Acetate Ophthalmic Suspension 1% for the Treatment of Inflammation Following Cataract Surgery in Children 0 to 3 Years of Age
Brief Title: KPI-121 1% Versus Prednisolone for the Treatment of Inflammation Following Cataract Surgery in Children
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: NDA #210565 did not trigger the need for a Pediatric Research Equity Act study.
Sponsor: Kala Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KPI-121-C-010
Record Dates: First submitted 2018-07-12; First posted 2018-07-24 (Actual); Results first posted 2020-04-07 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Ocular Inflammation
MeSH Terms: interventions — prednisolone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KPI-121 1% BID (twice daily) (Experimental)
  Interventions: Drug: KPI-121 1%
- Prednisolone acetate QID (four times daily) (Active Comparator)
  Interventions: Drug: Prednisolone acetate

INTERVENTIONS:
Drug: KPI-121 1% — eye drops
  Arms: KPI-121 1% BID (twice daily)
Drug: Prednisolone acetate — eye drops
  Other Names: Pred Forte
  Arms: Prednisolone acetate QID (four times daily)

SUMMARY:
This study is designed to assess how KPI-121 1% compares to prednisolone acetate in reducing inflammation after cataract surgery in young children. Approximately half the participants will receive KPI-121 1% eye drops and the other half will receive prednisolone acetate.

ELIGIBILITY:
Inclusion Criteria:

* Be a candidate for routine, uncomplicated cataract surgery

Exclusion Criteria:

* Have a post-traumatic cataract.
* Have suspected permanent low vision or blindness in the fellow non-study eye.
* Have active uveitis in either eye.
* Have an ocular neoplasm in either eye.
* Have the presence of viral, bacterial, or fungal disease in either eye.
* Have glaucoma, ocular hypertension, steroid-induced IOP (intraocular pressure) rise or elevated IOP

Max Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Byers Eye Institute at Stanford University, Palo Alto, California
  - Children's Eye Care, PC, Detroit, Michigan
  - Pediatric Ophthalmology of Erie, Inc., Erie, Pennsylvania
  - Houston Eye Associates, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- KPI-121 1% BID (Twice Daily): Subjects randomized to KPI-121 1% eye drops
- Prednisolone Acetate QID (Four Times Daily): Subjects randomized to Prednisolone acetate eye drops
Period: Overall Study
Arm/Group | KPI-121 1% BID (Twice Daily) | Prednisolone Acetate QID (Four Times Daily)
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KPI-121 1% BID (Twice Daily) | Prednisolone Acetate QID (Four Times Daily) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Continuous [Mean (Full Range); unit: months] | 44.0 [44 to 44] | 6.0 [6 to 6] | 25.0 [6 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Study Eye OD (right eye) [Number; unit: participants] | 1 | 1 | 2
Study Eye OS (left eye) [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Anterior Chamber Cell Grade
Description: Anterior chamber cell grading is a way of quantifying the amount of inflammation in inflammatory eye processes. Higher values indicate greater inflammation. The anterior chamber cell grading uses whole numbers from 0 (no cells) to 4 (> 30 cells) as follows:
  Anterior chamber cell grade 0 = no cells seen Anterior chamber cell grade 1 = 1 - 5 cells Anterior chamber cell grade 2 = 6 - 15 cells Anterior chamber cell grade 4 = greater than 30 cells
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Groups:
- KPI-121 1% BID: KPI-121 1%: eye drops
- Prednisolone Acetate QID: Prednisolone acetate: eye drops
Arm/Group | KPI-121 1% BID | Prednisolone Acetate QID
Number analyzed (Participants) | 1 | 1
Participants
  Anterior chamber cell grade = 0 | 0 | 0
  Anterior chamber cell grade = 1 | 1 | 1
  Anterior chamber cell grade = 2 | 0 | 0
  Anterior chamber cell grade = 3 | 0 | 0
  Anterior chamber cell grade = 4 | 0 | 0

2. Secondary Outcome: Modified Global Overall Assessment of Postoperative Inflammation
Description: The Modified Global Overall Assessment is a way of quantifying the amount of post operative healing that has occurred. Lower values indicate greater healing.The Modified Global Assessment grading uses whole numbers from 0 (clear) to 2 (not improving or worsening) as follows:
  0 = clear
  1. = improving satisfactorily
  2. = not improving or worsening
Time Frame: Day 15
Measure: Count of Participants; unit: Participants
Arm/Group | KPI-121 1% BID | Prednisolone Acetate QID
Number analyzed (Participants) | 1 | 1
Participants
  Modified Global Overall Assessment = 0 | 0 | 0
  Modified Global Overall Assessment = 1 | 1 | 1
  Modified Global Overall Assessment = 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of Investigational Product use at Visit 2 through conclusion of Visit 6, approximately 36 days.
Arm/Group | KPI-121 1% BID | Prednisolone Acetate QID
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KPI-121 1% BID (N=1) | Prednisolone Acetate QID (N=1)
Suture Related Complication (Eye disorders) | 1 (1) | 0 (0)
Increased Ocular Inflammation (Eye disorders) | 1 (1) | 0 (0)
Otitis Media (Ear and labyrinth disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Due to stopping the study after just two subjects were enrolled, no meaningful conclusions could be reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-11): https://cdn.clinicaltrials.gov/large-docs/23/NCT03596723/Prot_SAP_003.pdf